CLINICAL TRIAL: NCT00774397
Title: Antiviral Effect, Safety and Pharmacokinetics of BI 201335 NA in Hepatitis C Virus Genotype 1 Infected Treatment-naïve and Treatment-experienced Patients for 24 Weeks as Combination Therapy With Pegylated Interferon-alpha 2a and Ribavirin (Double-blinded, Randomised, Placebo-controlled, Phase II)
Brief Title: Antiviral Effect, Safety, and Pharmacokinetics of BI201335 +PegIFN/RBV in HCV-GT1 (SILEN-C1&2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.5; 2008-003538-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — faldaprevir; BID protein, human

ARMS (7):
- 240 mg QD TN (Experimental): 240 mg BI 201335 NA (Faldaprevir) once daily (QD) combined with PegIFN/RBV for 24 weeks, success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  Interventions: Drug: BI 201335 NA 240 mg QD; Drug: PegIFN/RBV
- 240 mg QD / LI-TN (Experimental): 240 mg BI 201335 NA (Faldaprevir) once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 (Faldaprevir) three days after first administration of PegIFN/RBV), success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  Interventions: Drug: BI 201335 NA 240 mg QD / LI; Drug: PegIFN/RBV
- Placebo (Placebo Comparator): Placebo once daily combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  Interventions: Drug: PegIFN/RBV; Drug: Placebo
- 120 mg QD / LI-TN (Experimental): 120 mg BI 201335 NA (Faldaprevir) once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in (LI) phase of PegIFN/RBV (i.e. initiation of BI 201335 (Faldaprevir) three days after first administration of PegIFN/RBV), followed by an additional 24 weeks of PegIFN/RBV in treatment naive (TN) patients
  Interventions: Drug: BI 201335 NA 120mg QD / LI; Drug: PegIFN/RBV
- 240 mg QD TE (Experimental): 240 mg BI 201335 NA (Faldaprevir) once daily (QD) combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV in treatment experienced (TE) patients
  Interventions: Drug: BI 201335 NA 240 mg QD; Drug: PegIFN/RBV
- 240 mg QD / LI-TE (Experimental): 240 mg BI 201335 NA (Faldaprevir) once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 (Faldaprevir) three days after first administration of PegIFN/RBV), success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-experienced (TE) patients
  Interventions: Drug: PegIFN/RBV; Drug: BI 201335 NA 240 mg QD
- 240 mg BID / LI-TE (Experimental): 240mg BI 201335 NA (Faldaprevir) twice daily combined with PegIFN/RBV for 24 or 48 weeks, with 3-day lead-in phase of PegIFN/RBV, in treatment-experienced patients
  Interventions: Drug: BI 201335 NA 240 mg BID; Drug: PegIFN/RBV

INTERVENTIONS:
Drug: BI 201335 NA 240 mg QD / LI — 240mg BI 201335 NA (Faldaprevir) once daily with a 3 days lead-in phase of PegIFN/RB, 24 weeks
  Other Names: Faldaprevir
  Arms: 240 mg QD / LI-TN
Drug: PegIFN/RBV — PegIFN (180 µg/wk) and RBV (1000/1200mg/d), 24 or 48 weeks
  Arms: 240 mg QD / LI-TN
Drug: BI 201335 NA 120mg QD / LI — 120mg BI 201335 NA (Faldaprevir) once daily, for 24 weeks
  Other Names: Faldaprevir
  Arms: 120 mg QD / LI-TN
Drug: PegIFN/RBV — PegIFN (180 µg/wk) and RBV (1000/1200mg/d),48 weeks
  Arms: 120 mg QD / LI-TN
Drug: BI 201335 NA 240 mg QD — 240mg BI 201335 NA (Faldaprevir) once daily, 24 weeks
  Other Names: Faldaprevir
  Arms: 240 mg QD TN
Drug: PegIFN/RBV — PegIFN (180 µg/wk) and RBV (1000/1200mg/d),48 weeks
  Arms: 240 mg QD TN
Drug: BI 201335 NA 240 mg QD — 240mg BI 201335 NA (Faldaprevir) once daily, 24 weeks
  Other Names: Faldaprevir
  Arms: 240 mg QD TE
Drug: PegIFN/RBV — PegIFN (180 µg/wk) and RBV (1000/1200mg/d), 24 or 48 weeks
  Arms: 240 mg QD TE
Drug: BI 201335 NA 240 mg BID — 240mg BI 201335 NA (Faldaprevir) twice, 24 weeks
  Other Names: Faldaprevir
  Arms: 240 mg BID / LI-TE
Drug: PegIFN/RBV — PegIFN (180 µg/wk) and RBV (1000/1200mg/d),48 weeks
  Arms: 240 mg BID / LI-TE
Drug: PegIFN/RBV — PegIFN (180 µg/wk) and RBV (1000/1200mg/d),48 weeks
  Arms: 240 mg QD / LI-TE
Drug: BI 201335 NA 240 mg QD — 240mg BI 201335 NA (Faldaprevir) once daily, 24 weeks
  Other Names: Faldaprevir
  Arms: 240 mg QD / LI-TE
Drug: PegIFN/RBV — PegIFN (180 µg/wk) and RBV (1000/1200mg/d), 24 or 48 weeks
  Arms: Placebo
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective was to investigate the antiviral effect, safety, and pharmacokinetics of BI 201335 (Faldaprevir), given as a soft gelatine capsule, in patients with hepatitis C virus (HCV) genotype 1 infection. Combination therapy of BI 201335 (Faldaprevir) with pegylated interferon α-2a (PegIFN) and ribavirin (RBV), with or without a 3-day lead-in, was assessed in treatment-naïve (TN) and treatment experienced (TE) patients.

ELIGIBILITY:
Inclusion criteria:

chronic HCV GT1; therapy-naive to IFN, PegIFN, or RBV; HCV VL >=100,000 IU/mL Liver biopsy within 2 years prior to study enrolment showing necroinflammatory activity or presence of fibrosis Normal retinal finding on fundoscopy within 6 months prior to Day 1 age 18-65 years Females and males with adequate contraception

Exclusion criteria:

Mixed genotype (1/2, 1/3, or 1/4), diagnosed by genotypic testing at screening Previous treatment with protease inhibitor Evidence of liver disease due to causes other than chronic HCV infection HIV-1 or HIV-2 positive HBV positive Decompensated liver disease, or history of decompensated liver disease Active or suspected malignancy or history of malignancy within the last 5 years History of alcohol or drug abuse within the past 12 months. Usage of any investigational drug within 30 days prior to enrolment, or 5 half-lives, whichever is longer Known hypersensitivity to any ingredient of the study drugs Condition that is defined as one which in the opinion of the investigator may put the patient at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study Alpha-fetoprotein value > 100ng/mL at screening; if >20ng/mL and <=100ng/mL, patients can be included if there is no evidence of liver cancer in two congruent imaging studies Total bilirubin > 1.5x ULN wiht ratio of direct/indirect >1. ALT or AST levels > 5x ULN INR prolonged to >1.5x ULN Exclusion criteria related to PegIFN and/or RBV restrictions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (100):
- United States (10):
  - 1220.5.0001 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1220.5.0008 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1220.5.0005 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1220.5.0006 Boehringer Ingelheim Investigational Site, Lutherville, Maryland
  - 1220.5.0002 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.5.0003 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.5.0007 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1220.5.0010 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 1220.5.0009 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1220.5.0004 Boehringer Ingelheim Investigational Site, Austin, Texas
- Argentina (5):
  - 1220.5.5401 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1220.5.5403 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1220.5.5405 Boehringer Ingelheim Investigational Site, Derqui, Pilar
  - 1220.5.5402 Boehringer Ingelheim Investigational Site, Rosario
  - 1220.5.5406 Boehringer Ingelheim Investigational Site, Rosario
- Australia (9):
  - 1220.5.6110 Boehringer Ingelheim Investigational Site, Camperdown, New South Wales
  - 1220.5.6109 Boehringer Ingelheim Investigational Site, Kogarah, New South Wales
  - 1220.5.6105 Boehringer Ingelheim Investigational Site, Randwick, New South Wales
  - 1220.5.6101 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 1220.5.6103 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 1220.5.6104 Boehringer Ingelheim Investigational Site, Woolloongabba, Queensland
  - 1220.5.6102 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1220.5.6107 Boehringer Ingelheim Investigational Site, Fitzroy, Victoria
  - 1220.5.6108 Boehringer Ingelheim Investigational Site, Parkville, Victoria
- Austria (3):
  - 1220.5.4303 Boehringer Ingelheim Investigational Site, Linz
  - 1220.5.4301 Boehringer Ingelheim Investigational Site, Vienna
  - 1220.5.4302 Boehringer Ingelheim Investigational Site, Vienna
- Canada (6):
  - 1220.5.1003 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1220.5.1007 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.5.1006 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1220.5.1001 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1220.5.1002 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1220.5.1004 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Czechia (2):
  - 1220.5.4202 Boehringer Ingelheim Investigational Site, Mělník
  - 1220.5.4203 Boehringer Ingelheim Investigational Site, Opava
- France (9):
  - 1220.5.3301A Boehringer Ingelheim Investigational Site, Clichy
  - 1220.5.3307A Boehringer Ingelheim Investigational Site, Créteil
  - 1220.5.3309A Boehringer Ingelheim Investigational Site, Lyon
  - 1220.5.3304A Boehringer Ingelheim Investigational Site, Marseille
  - 1220.5.3306A Boehringer Ingelheim Investigational Site, Montpellier
  - 1220.5.3302A Boehringer Ingelheim Investigational Site, Paris
  - 1220.5.3303A Boehringer Ingelheim Investigational Site, Paris
  - 1220.5.3308A Boehringer Ingelheim Investigational Site, Paris
  - 1220.5.3305A Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (14):
  - 1220.5.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.5.4903 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.5.4917 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.5.4914 Boehringer Ingelheim Investigational Site, Bochum
  - 1220.5.4913 Boehringer Ingelheim Investigational Site, Bonn
  - 1220.5.4915 Boehringer Ingelheim Investigational Site, Dortmund
  - 1220.5.4905 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.5.4912 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.5.4906 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1220.5.4908 Boehringer Ingelheim Investigational Site, Hamburg
  - 1220.5.4904 Boehringer Ingelheim Investigational Site, Hanover
  - 1220.5.4910 Boehringer Ingelheim Investigational Site, Leipzig
  - 1220.5.4909 Boehringer Ingelheim Investigational Site, Mainz
  - 1220.5.4907 Boehringer Ingelheim Investigational Site, Tübingen
- Netherlands (2):
  - 1220.5.3101 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1220.5.3102 Boehringer Ingelheim Investigational Site, Leiden
- Portugal (6):
  - 1220.5.3501 Boehringer Ingelheim Investigational Site, Coimbra
  - 1220.5.3504 Boehringer Ingelheim Investigational Site, Coimbra
  - 1220.5.3502 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.5.3503 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.5.3506 Boehringer Ingelheim Investigational Site, Porto
  - 1220.5.3507 Boehringer Ingelheim Investigational Site, Porto
- Romania (4):
  - 1220.5.4001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.5.4002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.5.4003 Boehringer Ingelheim Investigational Site, Bucharest
  - 1220.5.4004 Boehringer Ingelheim Investigational Site, Bucharest
- South Korea (11):
  - 1220.5.8210 Boehringer Ingelheim Investigational Site, Busan
  - 1220.5.8205 Boehringer Ingelheim Investigational Site, Daegu
  - 1220.5.8201 Boehringer Ingelheim Investigational Site, Pusan
  - 1220.5.8202 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.5.8206 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.5.8207 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.5.8208 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.5.8204 Boehringer Ingelheim Investigational Site, Seoungnam
  - 1220.5.8203 Boehringer Ingelheim Investigational Site, Sungnam
  - 1220.5.8209 Boehringer Ingelheim Investigational Site, Suwon
  - 1220.5.8211 Boehringer Ingelheim Investigational Site, Yangsan
- Spain (6):
  - 1220.5.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.5.3405 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.5.3401 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.5.3403 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.5.3404 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.5.3406 Boehringer Ingelheim Investigational Site, Madrid
- Switzerland (5):
  - 1220.5.4104 Boehringer Ingelheim Investigational Site, Bern
  - 1220.5.4102 Boehringer Ingelheim Investigational Site, La Chaux-de-Fonds
  - 1220.5.4103 Boehringer Ingelheim Investigational Site, Lugano
  - 1220.5.4101 Boehringer Ingelheim Investigational Site, Zurich
  - 1220.5.4106 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (8):
  - 1220.5.4405 Boehringer Ingelheim Investigational Site, Bristol
  - 1220.5.4401 Boehringer Ingelheim Investigational Site, London
  - 1220.5.4402 Boehringer Ingelheim Investigational Site, London
  - 1220.5.4406 Boehringer Ingelheim Investigational Site, London
  - 1220.5.4409 Boehringer Ingelheim Investigational Site, London
  - 1220.5.4410 Boehringer Ingelheim Investigational Site, London
  - 1220.5.4408 Boehringer Ingelheim Investigational Site, Nottingham
  - 1220.5.4403 Boehringer Ingelheim Investigational Site, Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-TN: Placebo once daily combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  [PegIFN/RBV (Pegylated interferon α-2a (Pegasys®)/ Ribavirin (Copegus®)): PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 120 mg QD / LI-TN: 120 mg BI 201335 (Faldaprevir) once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in (LI) phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), followed by an additional 24 weeks of PegIFN/RBV in treatment naive (TN) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240 mg QD / LI-TN: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240 mg QD-TN: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240 mg QD / LI-TE: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-experienced (TE) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240 mg QD-TE: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV in treatment experienced (TE) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240 mg BID / LI-TE: 240 mg BI 201335 twice daily (BID) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), followed by an additional 24 weeks of PegIFN/RBV in treatment experienced (TE) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
Period: Overall Study
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Started | 71 | 69 | 143 | 146 | 143 | 76 | 71
Completed | 57 | 56 | 113 | 129 | 97 | 54 | 41
Not Completed | 14 | 13 | 30 | 17 | 46 | 22 | 30
Not completed — Adverse Event | 1 | 3 | 16 | 8 | 8 | 3 | 16
Not completed — Lack of Efficacy | 11 | 4 | 5 | 3 | 27 | 15 | 9
Not completed — Protocol Violation | 0 | 1 | 3 | 1 | 2 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 1 | 0
Not completed — Refused to continue trial medication | 1 | 3 | 2 | 2 | 6 | 2 | 3
Not completed — Not treated | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other than those stated above | 1 | 1 | 3 | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set: The treated set (TS) included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment, whether randomised or not
Groups:
- Placebo-TN: Placebo once daily combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  [PegIFN/RBV : PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- Total: Total of all reporting groups
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE | Total
Number analyzed (Participants) | 71 | 69 | 143 | 146 | 142 | 76 | 70 | 717
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (10.86) | 46.3 (10.92) | 44.7 (10.18) | 46.3 (10.48) | 48.7 (9.58) | 49.6 (8.42) | 50.1 (8.34) | 47.14 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 69 | 67 | 41 | 26 | 29 | 291
  Male | 41 | 40 | 74 | 79 | 101 | 50 | 41 | 426

OUTCOME MEASURES:

1. Primary Outcome: Virological Response 4 Weeks After the End of Treatment With BI 201335 or Placebo
Description: An achieved virological response is defined as the plasma Hepatitis C Virus RiboNucleic Acid (HCV RNA) level below the lower limit of detection (BLD).
  This data was only collected for patients, who stopped trial participation at Week 24 and did not continue with PegIFN/RBV until Week 48.
  The lower limit of quantification (BLQ) of this assay was 25 IU/mL and the lower limit of detection (BLD) was 10 IU/mL at the time of the protocol finalisation. During the course of the trial, the manufacturer defined BLD as '< 25 IU/mL, not detectable' and BLQ as '< 25 IU/mL, detectable'.
Time Frame: Week 28
Population: Per protocol set (PPS): PPS was subset of full analysis set,consisted of all patients without important protocol deviations .
  FAS was composed of all randomised patients who took at least 1 dose of study medication.
  For this outcome, only patients who were not on PegIFN/RBV treatment 4 weeks after stop of BI 201335 or Placebo were investigated.
Measure: Number; unit: percentage of patients
Groups:
- Placebo-TN: Placebo once daily combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 13 | 14 | 77 | 72 | 88 | 30 | 27
percentage of patients | 0.0 | 14.3 | 59.7 | 75.0 | 20.5 | 3.3 | 0.0

2. Primary Outcome: Sustained Virological Response 24 Weeks (SVR24) After Completion of All Therapy
Description: Virological (VL) response was defined as the plasma HCV RNA level below the lower limit of detection.
  The first VL measurement that occurred in the time window ≥ Day 155 (from End Of Treatment on) was selected for the determination of SVR24.
  Therefore, patients with virological load BLD 24 weeks after completion of therapy, who had a rebound after this time point (outside the defined time window of 155 days after end of all treatments) were identified as SVR24 achieved.
Time Frame: Day 155 after the end of all treatment
Population: Per protocol set
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 56.3 [44.7 to 67.3] | 72.5 [60.9 to 81.6] | 72.3 [64.4 to 79.1] | 83.8 [76.9 to 88.9] | 28.2 [21.4 to 36.1] | 40.8 [30.4 to 52.1] | 31.4 [21.8 to 43.1]
Statistical Analysis 1: Comparison: Placebo-TN vs 120 mg QD / LI-TN; Test type: Superiority or Other; p = 0.0537, Fisher Exact — P-value based on Fisher's exact test (2-sided)
Statistical Analysis 2: Comparison: Placebo-TN vs 240 mg QD / LI-TN; Test type: Superiority or Other; p = 0.0213, Fisher Exact — P-value based on Fisher's exact test (2-sided)
Statistical Analysis 3: Comparison: Placebo-TN vs 240 mg QD-TN; Test type: Superiority or Other; p < 0.0001, Fisher Exact — P-value based on Fisher's exact test (2-sided)
Statistical Analysis 4: Comparison: 240 mg QD / LI-TE; Test type: Superiority or Other; p < 0.0001, Fisher Exact — P-value based on Fisher's exact test (2-sided)
Statistical Analysis 5: Comparison: 240 mg QD-TE; Test type: Superiority or Other; p < 0.0001, Fisher Exact — P-value based on Fisher's exact test (2-sided)
Statistical Analysis 6: Comparison: 240 mg BID / LI-TE; Test type: Superiority or Other; p < 0.0001, Fisher Exact — P-value based on Fisher's exact test (2-sided)

3. Secondary Outcome: Virological Response at Week 2
Description: Viral load (plasma HCV RNA level) below the lower limit of quantification at Week 2 (< 25 IU/ml, detectable or undetectable)
Time Frame: Week 2
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 1.4 | 69.6 | 66.7 | 82.4 | 27.5 | 34.2 | 47.1

4. Secondary Outcome: Virological Response at Week 4
Description: Viral load (plasma HCV RNA level) below the lower limit of quantification at Week 4 (< 25 IU/ml, detectable or undetectable)
Time Frame: Week 4
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 16.9 | 89.9 | 86.5 | 93.7 | 63.4 | 60.5 | 68.6

5. Secondary Outcome: Early Virological Response (EVR)
Description: Early Virological Response (EVR) is defined as ≥ 2 log 10 reduction in plasma HCV RNA level from baseline at Week 12
Time Frame: Baseline and Week 12
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 84.5 | 89.9 | 88.7 | 93.0 | 72.5 | 76.3 | 62.9

6. Secondary Outcome: Extended Rapid Virological Response (eRVR)
Description: Extended Rapid Virological Response (eRVR) is defined as plasma HCV RNA levels below the lower limit of quantification at Week 4 and below the lower limit of detection at Week 12
Time Frame: Week 4 and Week 12
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 15.5 | 85.5 | 80.9 | 90.8 | 52.1 | 52.6 | 51.4

7. Secondary Outcome: Complete Early Virological Response (cEVR)
Description: Complete Early Virological Response (cEVR) is defined as plasma HCV RNA level below the lower limit of detection at Week 12
Time Frame: Week 12
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 42.3 | 87.0 | 84.4 | 93.0 | 58.5 | 59.2 | 52.9

8. Secondary Outcome: End of Treatment Response at Week 24
Description: End of Treatment Response of BI 201335 or placebo (ETR BI 201335/placebo ) is defined as plasma HCV RNA level below the lower limit of detection at Week 24.
Time Frame: Week 24
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 73.2 | 82.6 | 77.3 | 88.0 | 58.5 | 52.6 | 52.9

9. Secondary Outcome: End of Treatment Response at End of All Therapy
Description: End of Treatment Response (ETR) is defined as plasma HCV RNA level below the lower limit of detection at end of all therapy, i.e. at Week 24 or Week 48
Time Frame: Week 24 or Week 48
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 69.0 | 72.5 | 78.0 | 81.7 | 48.6 | 46.1 | 45.7

10. Secondary Outcome: Sustained Virological Response 12 Weeks (SVR12) After Completion of All Therapy
Description: Sustained Virological Response 12 Weeks (SVR12) after completion of all therapy is defined as plasma HCV RNA level below the lower limit of detection at 12 weeks after completion of all therapy, i.e. at Week 36 or 60
Time Frame: Week 36 or Week 60
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 50.7 | 68.1 | 65.2 | 74.6 | 26.1 | 35.5 | 27.1

11. Secondary Outcome: Time to Reach a Plasma HCV RNA Level Below the Lower Limit of Detection
Description: Summary of time (i.e Median number of days) to reach a plasma HCV RNA level below limit of detection (BLD)
Time Frame: On or after day 155 post end of all treatment
Population: Per protocol set
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
Days | 113 [29 to 197] | 29 [8 to 113] | 29 [4 to 113] | 29 [4 to 113] | 56 [8 to 143] | 56 [8 to 169] | 29 [15 to 143]

12. Secondary Outcome: Time to Loss of Virological Response
Description: Time to loss of virological response, defined as the last value below the lower limit of detection in a patient who subsequently had 2 consecutive plasma HCV RNA level measurements ≥100 IU/mL. Patients that did not achieve suppression of plasma HCV RNA levels below the lower limit of detection until Week 24 were defined as having a time to failure of zero.
  Time is expressed in Median number of days.
Time Frame: Week 24
Population: Per protocol set
Measure: Median (95% Confidence Interval); unit: Number of days
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 57 | 64 | 128 | 138 | 100 | 50 | 48
Number of days | NA [NA to NA] — More than 50% of all patients of the respective group have no loss of virological response at all, therefore no median can be calculated | NA [NA to NA] — More than 50% of all patients of the respective group have no loss of virological response at all, therefore no median can be calculated | NA [NA to NA] — More than 50% of all patients of the respective group have no loss of virological response at all, therefore no median can be calculated | NA [NA to NA] — More than 50% of all patients of the respective group have no loss of virological response at all, therefore no median can be calculated | 230 [0 to NA] — NA stands for infinity | 370 [0 to NA] — NA stands for infinity | 370 [0 to NA] — NA stands for infinity

13. Secondary Outcome: Virological Rebound
Description: Virological rebound is defined as increase of ≥ 1 log 10 in plasma HCV RNA level from a quantifiable nadir, or to ≥ 250 IU/mL after previous nadir < 25 IU/mL (detectable), or to ≥ 100 IU/mL after a previous viral load below the lower limit of detection.
  Note that this is numerical rebound, not requiring confirmation with a re-measurement.
Time Frame: Week 24 or Week 48
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 28.2 | 17.4 | 19.9 | 12.0 | 67.6 | 53.9 | 60.0

14. Secondary Outcome: Breakthrough on BI 201335/Placebo (Rebound While All 3 Treatments Were Still Ongoing)
Description: Number of patients with Unconfirmed rebound ( ≥ 1log10 increase in HCV mRNA) while on BI201335/placebo + 5 days washout.
Time Frame: Up to Week 24
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 4.2 | 5.8 | 5.0 | 3.5 | 25.4 | 28.9 | 17.1

15. Secondary Outcome: Breakthrough on PegIFN/RBV (Rebound While Only PegIFN/RBV Treatment Alone Was Still Ongoing)
Description: Number of patients with Unconfirmed rebound (≥ 1log10 increase in HCV mRNA) while on PegIFN/RBV treatment + 5 days washout.
Time Frame: Week 24 through Week 48
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 4.2 | 2.9 | 0.7 | 0.0 | 4.9 | 6.6 | 7.1

16. Secondary Outcome: Relapse
Description: Relapse was rebound after the viral load at end of all treatment had been below the lower limit of detection, or, if the value at end of all treatment was missing, after both the last value before End of Treatment (EOT) and the first value after End of Treatment were below the lower limit of detection.
  Patients could experience relapse at any point post-treatment.
Time Frame: post-End of treatment (i.e. post 48 weeks)
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients | 15.5 | 7.2 | 10.6 | 7.7 | 26.8 | 11.8 | 20.0

17. Secondary Outcome: Change From Baseline to Week 24 in Diastolic Blood Pressure and Systolic Blood Pressure
Description: Baseline is defined as the last value before the initial drug administration of BI 201335 or placebo.
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with change from baseline in Systolic blood pressure and Diastolic blood pressure at Week 24)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 61 | 60 | 115 | 130 | 102 | 55 | 42
mmHg
  Diastolic Blood Pressure | -0.5 (9.11) | 0.8 (12.41) | -1.4 (10.87) | -1.9 (10.19) | -1.4 (9.34) | -1.8 (10.39) | -5.3 (10.27)
  Systolic Blood Pressure | -2.6 (11.48) | -3.8 (15.51) | -4.6 (14.59) | -3.2 (13.63) | -1.8 (14.21) | -3.4 (12.85) | -8.0 (14.38)

18. Secondary Outcome: Change From Baseline to Week 24 in Pulse Rate
Description: Baseline is defined as the last value before the administration of BI 201335 or placebo.
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with change from baseline in Pulse rate at Week 24)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 61 | 60 | 115 | 130 | 102 | 55 | 42
bpm | 4.1 (10.22) | 3.1 (11.37) | 4.1 (14.53) | 5.3 (11.45) | 5.5 (11.30) | 7.6 (10.77) | 3.1 (13.46)

19. Secondary Outcome: Change From Baseline to Week 24 in Weight of the Patients
Description: Baseline is defined as the last value before the administration of BI 201335 or placebo.
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with change from baseline in Weight at Week 24)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 61 | 60 | 115 | 130 | 101 | 55 | 42
kg | -3.3 (3.11) | -3.7 (3.14) | -4.2 (3.81) | -4.8 (5.07) | -3.4 (3.36) | -4.3 (3.67) | -4.8 (4.40)

20. Secondary Outcome: Global Assessment of Tolerability
Description: The investigator was to assess the tolerability of trial medication based on adverse events (AEs) and the laboratory evaluation.
  Tolerability was assessed by the investigator according to the categories 'good', 'satisfactory', 'not satisfactory', and 'bad'.
Time Frame: Week 24
Population: Per protocol set
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 141 | 142 | 142 | 76 | 70
percentage of patients
  Good | 46.5 | 40.6 | 41.1 | 47.2 | 41.5 | 31.6 | 20.0
  Satisfactory | 33.8 | 36.2 | 36.2 | 31.7 | 33.1 | 40.8 | 37.1
  Not satisfactory | 8.5 | 11.6 | 12.1 | 12.0 | 13.4 | 14.5 | 22.9
  Bad | 5.6 | 2.9 | 5.0 | 6.3 | 9.2 | 9.2 | 20.0
  Not assessable | 1.4 | 2.9 | 4.3 | 0.0 | 1.4 | 0.0 | 0.0
  Missing | 4.2 | 5.8 | 1.4 | 2.8 | 1.4 | 3.9 | 0.0

21. Secondary Outcome: Change From Baseline to Week 24 in Haemoglobin of the Patients
Description: Baseline is defined as the last value before the administration of BI 201335 or placebo.
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with change from baseline in Haemoglobin at Week 24)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 60 | 59 | 114 | 129 | 103 | 55 | 40
g/dL | -3.51 (1.526) | -3.41 (1.406) | -3.41 (1.177) | -3.43 (1.493) | -3.19 (1.447) | -3.41 (1.285) | -3.82 (1.997)

22. Secondary Outcome: Number of Patients [N(%)] With Transitions Relative to Reference Range for Laboratory Parameter Haemoglobin
Description: Number of patients with normal or high baseline moved to low .
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with normal or high baseline Haemoglobin)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 70 | 67 | 137 | 146 | 139 | 76 | 67
percentage of patients | 64.3 | 62.7 | 51.1 | 53.4 | 45.3 | 63.2 | 53.7

23. Secondary Outcome: Change From Baseline to Week 24 in Absolute Neutrophils of the Patients
Description: Baseline is defined as the last value before the administration of BI 201335 or placebo.
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with change from baseline in Absolute Neutrophils at Week 24)
Measure: Mean (Standard Deviation); unit: GI/L
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 58 | 58 | 111 | 129 | 102 | 55 | 39
GI/L | -2.57 (1.784) | -1.84 (1.497) | -1.83 (2.788) | -2.10 (1.551) | -1.87 (1.567) | -1.47 (1.680) | -1.84 (1.885)

24. Secondary Outcome: Number of Patients [N(%)] With Transitions Relative to Reference Range for Laboratory Parameter Absolute Neutrophils
Description: Number of patients with normal or high baseline moved to low .
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with normal or high baseline Absolute Neutrophils)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 68 | 65 | 134 | 139 | 126 | 66 | 57
percentage of patients | 70.6 | 66.2 | 47.8 | 45.3 | 50.0 | 54.5 | 47.4

25. Secondary Outcome: Change From Baseline to Week 24 in ALT/GPT,SGPT of the Patients
Description: Baseline is defined as the last value before the drug administration of BI 201335 or placebo.
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with change from baseline in ALT/GPT,SGPT at Week 24)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 60 | 60 | 116 | 130 | 102 | 55 | 42
U/L | -92.0 (86.98) | -67.7 (65.95) | -64.2 (80.46) | -70.2 (92.76) | -50.8 (77.43) | -62.0 (68.60) | -61.0 (80.46)

26. Secondary Outcome: Number of Patients [N(%)] With Transitions Relative to Reference Range for Laboratory Parameter ALT/GPT,SGPT
Description: Number of patients with normal or low baseline moved to high .
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with normal or low baseline ALT/GPT,SGPT)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 11 | 10 | 32 | 26 | 24 | 6 | 10
percentage of patients | 0.0 | 10.0 | 3.1 | 0.0 | 8.3 | 16.7 | 20.0

27. Secondary Outcome: Change From Baseline to Week 24 in Total Bilirubin of the Patients
Description: Baseline is defined as the last value before the administration of BI 201335 or placebo.
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with change from baseline in Total Bilirubin at Week 24)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 61 | 60 | 116 | 130 | 103 | 55 | 42
mg/dL | 0.03 (0.181) | 0.70 (0.625) | 1.65 (1.279) | 1.51 (0.983) | 1.37 (0.959) | 1.09 (0.996) | 3.04 (2.203)

28. Secondary Outcome: Number of Patients [N(%)] With Transitions Relative to Reference Range for Laboratory Parameter Total Bilirubin
Description: Number of patients with normal or low baseline moved to high .
Time Frame: Baseline and Week 24
Population: Treated Set (for patients with normal or low baseline Total Bilirubin)
Measure: Number; unit: percentage of patients
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 69 | 66 | 132 | 146 | 136 | 74 | 68
percentage of patients | 0.0 | 9.1 | 15.9 | 8.9 | 29.4 | 17.6 | 33.8

29. Secondary Outcome: Trough Concentration (Cpre,ss) of Faldaprevir at Steady State
Description: C(pre,ss) is defined as pre-dose (trough) concentration of Faldaprevir in plasma at steady state immediately before administration of the next dose.
Time Frame: Week 8, week 10, week 12, week 24
Population: All evaluable patients were included in the pharmacokinetic analysis. A patient was considered to be not evaluable if the patient had a protocol violation relevant to the evaluation of pharmacokinetics or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 69 | 143 | 146 | 142 | 76 | 70
ng/mL
  week 8(N=52,108,116,107,47,32) | 1310 (81.7) | 6550 (106) | 6190 (169) | 7230 (94.3) | 6410 (95.4) | 51100 (55.1)
  week 10(N=54,98,101,94,54,29) | 1220 (91.3) | 6530 (118) | 6340 (99.7) | 6370 (137) | 7020 (108) | 43500 (72.2)
  week 12(N=53,113,119,105,56,30) | 1240 (91.1) | 6380 (125) | 6780 (100) | 6400 (123) | 5980 (91.2) | 46300 (58.7)
  week 24(N=47,86,95,78,39,26) | 1170 (142) | 6440 (109) | 6610 (132) | 6630 (102) | 4280 (179) | 33900 (509)

30. Secondary Outcome: Trough Concentration (Cpre,ss) of Ribavirin at Steady State (Receiving 1000 mg/Day RBV)
Description: C(pre,ss) is defined as pre-dose (trough) concentration of Ribavirin in plasma at steady state immediately before administration of the next dose.
Time Frame: Week 8, week 10, week 12, week 24
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 143 | 146 | 142 | 76 | 70
ng/mL
  week 8(N=23,25,46,43,38,20,12) | 2260 (26.6) | 1920 (37.9) | 2320 (30.8) | 2200 (28.7) | 2150 (26.4) | 2090 (26.0) | 2180 (27.1)
  week 10(N=22,27,50,38,34,25,11) | 2210 (28.2) | 1960 (33.3) | 2290 (30.8) | 2330 (23.8) | 2190 (28.9) | 2140 (24.6) | 2300 (21.5)
  week 12(N=22,27,45,47,37,21,11) | 2200 (25.1) | 2060 (35.9) | 2290 (33.6) | 2340 (29.5) | 2140 (28.2) | 2150 (23.6) | 2300 (27.3)
  week 24(N=21,18,37,34,28,16,11) | 2370 (34.6) | 2100 (45.3) | 2390 (29.6) | 2260 (37.3) | 1960 (35.5) | 2270 (25.0) | 1970 (47.1)

31. Secondary Outcome: Trough Concentration (Cpre,ss) of Ribavirin at Steady State (Receiving 1200 mg/Day RBV)
Description: as for outcome 30
Time Frame: Week 8, week 10, week 12, week 24
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 143 | 146 | 142 | 76 | 70
ng/mL
  week 8(N=24,21,45,48,49,25,23) | 1670 (118) | 2010 (30.4) | 2060 (26.5) | 2170 (30.4) | 2060 (30.5) | 2170 (40.2) | 1880 (37.2)
  week 10(N=27,22,43,45,47,22,22) | 1780 (97.3) | 1970 (28.5) | 2100 (26.1) | 2280 (26.5) | 2090 (30.5) | 1980 (35.3) | 2090 (34.4)
  week 12(N=27,21,46,47,44,25,22) | 1880 (59.1) | 1900 (37.0) | 2090 (21.7) | 2260 (26.0) | 2190 (29.0) | 2010 (33.2) | 1950 (24.9)
  week 24(N=21,19,33,39,38,18,17) | 2030 (27.0) | 2390 (23.3) | 1970 (32.2) | 2250 (23.0) | 2180 (27.7) | 2050 (31.9) | 2220 (29.7)

32. Secondary Outcome: Trough Concentration (Cpre,ss) of PegIFN at Steady State
Description: C(pre,ss) is defined as pre-dose (trough) concentration of PegIFN in plasma at steady state immediately before administration of the next dose.
Time Frame: Week 8, week 10, week 12, week 24
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo-TN | 120 mg QD / LI-TN | 240 mg QD / LI-TN | 240 mg QD-TN | 240 mg QD / LI-TE | 240 mg QD-TE | 240 mg BID / LI-TE
Number analyzed (Participants) | 71 | 69 | 143 | 146 | 142 | 76 | 70
ng/mL
  week 8(N=55,46,80,91,80,36,33) | 14500 (83.9) | 14800 (59.9) | 14900 (41.1) | 15100 (58.5) | 11300 (151) | 11100 (125) | 12300 (95.1)
  week 10(N=46,48,88,94,80,40,33) | 14700 (86.6) | 13400 (87.1) | 14600 (70.2) | 15500 (52.2) | 11300 (144) | 11600 (155) | 12500 (85.4)
  week 12(N=54,51,100,107,105,56,42) | 15600 (77.9) | 13000 (102) | 13700 (89.4) | 14600 (70.5) | 13100 (105) | 13800 (110) | 13500 (102)
  week 24(N=49,42,74,87,75,40,38) | 17300 (45.4) | 17200 (83.8) | 16900 (42.2) | 16700 (50.3) | 15600 (44.0) | 15300 (63.3) | 15700 (38.5)

ADVERSE EVENTS:
Time Frame: Up to week 72 . Only SAEs related to the study drugs or study design (defined by the investigator) were to be reported from Week 72 up to Week 120.
Description: In the participant flow all randomised patients are counted with their randomised treatment. But for the AE analyses each patient is reported in that treatment which he has actually taken (which could be different from the treatment he was randomised to). In addition, only patients who take at least treatment once are included in the AE analyses.
Groups:
- 120mg QD/LI-TN: 120 mg BI 201335 (Faldaprevir) once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in (LI) phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), followed by an additional 24 weeks of PegIFN/RBV in treatment naive (TN) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240mg QD/LI-TN: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240mg QD-TN: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-naive (TN) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240mg QD/LI-TE: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), success-dependently followed by re-randomisation to stop or to an additional 24 weeks of PegIFN/RBV in treatment-experienced (TE) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240mg QD-TE: 240 mg BI 201335 once daily (QD) combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV in treatment experienced (TE) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
- 240mg BID/LI-TE: 240 mg BI 201335 twice daily (BID) combined with PegIFN/RBV for 24 weeks, with a 3-day lead-in phase of PegIFN/RBV (i.e. initiation of BI 201335 three days after first administration of PegIFN/RBV), followed by an additional 24 weeks of PegIFN/RBV in treatment experienced (TE) patients
  [PegIFN/RBV: PegIFN (180 µg/wk) and RBV (1000/1200mg/d)]
Arm/Group | Placebo-TN | 120mg QD/LI-TN | 240mg QD/LI-TN | 240mg QD-TN | 240mg QD/LI-TE | 240mg QD-TE | 240mg BID/LI-TE
Serious Adverse Events (participants affected / at risk) | 2/71 | 3/68 | 18/138 | 12/149 | 10/141 | 5/76 | 13/69
Other Adverse Events (participants affected / at risk) | 65/71 | 65/68 | 135/138 | 143/149 | 135/141 | 74/76 | 68/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-TN (N=71) | 120mg QD/LI-TN (N=68) | 240mg QD/LI-TN (N=138) | 240mg QD-TN (N=149) | 240mg QD/LI-TE (N=141) | 240mg QD-TE (N=76) | 240mg BID/LI-TE (N=69)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Microvascular angina (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cryoglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Superinfection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicectomy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-TN (N=71) | 120mg QD/LI-TN (N=68) | 240mg QD/LI-TN (N=138) | 240mg QD-TN (N=149) | 240mg QD/LI-TE (N=141) | 240mg QD-TE (N=76) | 240mg BID/LI-TE (N=69)
Anaemia (Blood and lymphatic system disorders) | 12 | 14 | 16 | 22 | 10 | 10 | 13
Neutropenia (Blood and lymphatic system disorders) | 8 | 9 | 11 | 9 | 7 | 10 | 3
Dry eye (Eye disorders) | 2 | 1 | 7 | 4 | 8 | 3 | 3
Ocular icterus (Eye disorders) | 1 | 1 | 8 | 2 | 2 | 8 | 6
Vision blurred (Eye disorders) | 0 | 2 | 4 | 2 | 7 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1 | 1 | 7 | 10 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 10 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 4 | 9 | 6 | 10 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 6 | 9 | 14 | 11 | 10 | 11
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 5 | 3 | 1 | 5
Constipation (Gastrointestinal disorders) | 1 | 5 | 6 | 3 | 7 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 13 | 9 | 44 | 40 | 45 | 24 | 26
Dry mouth (Gastrointestinal disorders) | 2 | 3 | 7 | 9 | 10 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 3 | 18 | 13 | 10 | 5 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 4 | 1 | 6 | 0 | 4
Nausea (Gastrointestinal disorders) | 14 | 17 | 65 | 66 | 68 | 40 | 43
Toothache (Gastrointestinal disorders) | 1 | 4 | 2 | 5 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 14 | 25 | 34 | 24 | 17 | 21
Asthenia (General disorders) | 15 | 10 | 33 | 41 | 34 | 15 | 19
Chills (General disorders) | 8 | 4 | 14 | 16 | 10 | 9 | 1
Fatigue (General disorders) | 24 | 19 | 32 | 39 | 49 | 30 | 25
Influenza like illness (General disorders) | 34 | 26 | 48 | 55 | 44 | 21 | 23
Injection site erythema (General disorders) | 7 | 3 | 7 | 9 | 8 | 1 | 3
Irritability (General disorders) | 10 | 8 | 15 | 13 | 27 | 12 | 7
Pyrexia (General disorders) | 11 | 10 | 26 | 30 | 25 | 12 | 16
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3 | 13 | 3 | 2 | 4 | 0
Jaundice (Hepatobiliary disorders) | 1 | 4 | 27 | 37 | 25 | 10 | 26
Herpes simplex (Infections and infestations) | 4 | 1 | 0 | 1 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 4 | 4 | 6 | 4 | 1 | 5
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 7 | 6 | 2 | 5
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 2 | 4
Haemoglobin decreased (Investigations) | 4 | 2 | 1 | 6 | 3 | 2 | 0
Weight decreased (Investigations) | 4 | 3 | 9 | 10 | 7 | 5 | 7
Decreased appetite (Metabolism and nutrition disorders) | 11 | 16 | 28 | 31 | 28 | 14 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 11 | 15 | 16 | 13 | 11 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 10 | 7 | 12 | 2 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 1 | 4 | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 6 | 9 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 14 | 26 | 35 | 24 | 17 | 17
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 1 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 4 | 2 | 1 | 2
Disturbance in attention (Nervous system disorders) | 3 | 2 | 5 | 2 | 8 | 3 | 3
Dizziness (Nervous system disorders) | 5 | 4 | 9 | 10 | 16 | 4 | 5
Dysgeusia (Nervous system disorders) | 0 | 3 | 4 | 2 | 8 | 3 | 5
Headache (Nervous system disorders) | 27 | 28 | 46 | 51 | 56 | 32 | 30
Lethargy (Nervous system disorders) | 5 | 3 | 5 | 3 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 1 | 2 | 0 | 3 | 1 | 4
Anxiety (Psychiatric disorders) | 3 | 3 | 5 | 6 | 11 | 4 | 2
Depressed mood (Psychiatric disorders) | 3 | 0 | 2 | 3 | 6 | 2 | 5
Depression (Psychiatric disorders) | 7 | 9 | 16 | 17 | 19 | 3 | 4
Insomnia (Psychiatric disorders) | 17 | 12 | 22 | 28 | 30 | 12 | 14
Mood swings (Psychiatric disorders) | 5 | 1 | 2 | 3 | 1 | 5 | 1
Sleep disorder (Psychiatric disorders) | 3 | 3 | 16 | 12 | 9 | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 22 | 18 | 25 | 13 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 13 | 13 | 24 | 7 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 8 | 8 | 6 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 16 | 29 | 23 | 17 | 9 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 16 | 25 | 22 | 26 | 13 | 20
Eczema (Skin and subcutaneous tissue disorders) | 3 | 4 | 9 | 7 | 4 | 5 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 8 | 9 | 6 | 6 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 1 | 7 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 13 | 14 | 19 | 10 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 22 | 49 | 56 | 43 | 34 | 23
Rash (Skin and subcutaneous tissue disorders) | 12 | 14 | 39 | 40 | 35 | 14 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.